CLINICAL TRIAL: NCT04116788
Title: Analysis and Reducing Modalities for Artefacts Generated by Bone Conduction Implants and Cochlear Implants Subjected to an MRI Magnetic Field - Artefact
Brief Title: Analysis and Reducing Modalities for Artefacts Generated by Bone Conduction Implants and Cochlear Implants Subjected to an MRI Magnetic Field
Acronym: Artefact
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Arnaud Devèze (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-A01036-45
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Hearing Implants; Implant Hearing Artefact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Artefact IRM assessment — IRM

SUMMARY:
Investigator team hypothesize that artifacts generated by the presence of an acoustic implant subjected to the magnetic field of the MRI are variable depending on the type of sequence and can be reduced by structural modifications of the implant and by variations in its appearance positioning with respect to the magnetic field MRI.

DETAILED DESCRIPTION:
Little scientific data is available on the artifacts generated by hearing implants. Indeed, hearing rehabilitation for deaf people was given priority over the potential constraints of imaging. Investigator team find less than 10 articles with a search of following keywords on the pubmed database: Artifacts AND MRI AND cochlear implants. Only one of these articles deals with demagnetization. There is only one article dealing with artifacts with the Bonebridge implant. There are no studies with the Attract implant and a recent one with the new Synchrony mobile magnet implant, but by removing the magnet which implies a minimum response time and therefore not compatible with emergency care.

In total, the literature is quite poor mainly considering the priority of auditory rehabilitation on the realization of subsequent imaging.

However, the current "democratization" of hearing implants and their increasing use in children and adults requires reflection on not only the safety of examinations of healthy volunteers, but also of the implant itself. also on the relevance of the interpretation of imaging especially cerebral.

The pilot study done, suggested that the placement of the implant (in this case the Bonebridge) has an influence on the size of the artifact and the possibilities of interpretation.

It seems appropriate to continue this protocol of analysis, both on the implants in bone conduction, and also on the cochlear implants to demonstrate the impact of the implant on the MRI images and also the impact of the magnetic field on the implant itself, and possibly publish recommendations for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* free of otological, neurological or psychiatric pathology
* absence of contraindication to MRI *
* free and informed consent signed

Exclusion Criteria:

* minor subject, major guardianship or trusteeship and major protected under the law (pregnant women, nursing, parturiante, persons deprived of their liberty)
* suject carrier of an implantable device or para magnetic
* contraindication to MRI *
* revious otological pathology, tinnitus, deafness
* revious cerebral pathology
* unable to understand the objectives, issues and risks of the study and to give free and informed consent.

  * Contraindications to MRI are:

Claustrophobia Anxiety attack Morphotype does not allow access to MRI

Wearing a metal implant, for example:

* a pacemaker
* ferromagnetic surgical clips
* foreign bodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Artefact surface ratio | 1 day
  The primary endpoint will be the percentage of artefact area (SA) induced by the magnetic implant relative to the overall sectional area of the artifactless skull section (SC).
  The measured artefact surface will therefore be related to the reference surface and the artefact percentage will be calculated by the following formula:
  Ratio (R) = Area artifact (SA) / Area cut (SC) * 100

CONTACTS AND LOCATIONS:
Locations (1):
- Clairval Private Hospital, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: Undecided